CLINICAL TRIAL: NCT04414852
Title: A Multi-center, Non-randomized, Open-label, Parallel Study to Evaluate the Pharmacokinetics of Apatinib Mesylate in Subjects With Impaired Renal Function and Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Apatinib in Subjects With Impaired Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR-APTN-I-011
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Subjects With Impaired Renal Function and Healthy Subjects
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild renal impairment (Experimental)
  Interventions: Drug: Apatinib Mesylate
- moderate remal impairment (Experimental)
  Interventions: Drug: Apatinib Mesylate
- normal renal impairment (Active Comparator)
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — All the subjects will be administrated with 250mg apatinib on day 1

SUMMARY:
The primary objective of the study is to compare the pharmacokinetics of apatinib in subjects with impaired renal function and healthy subjects, to give dose recommendations for patients with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

for subjects with impaired renal function

* Able to comprehend and willing to sign an informed consent form (ICF)
* 18-70 years of age.
* 19 kg/m2<BMI <19-28 kg/m2
* eGFR (MDRD equation) for mild impaired renal function: 60-89 mL/min/1.73 m2 eGFR (MDRD equation) for moderate impaired renal function: 30-59 mL/min/1.73 m2
* In good health, except for kidney disease and complications, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG;
* Agree to take approved method of contraception during the clinical trail and 8 weeks after the last dose of apatinib. Female subject should be negative in the pregnancy test;

for healthy subjects:

* Able to comprehend and willing to sign an informed consent form (ICF)
* 18-70 years of age.
* 19 kg/m2<BMI <19-28 kg/m2
* eGFR (MDRD equation) for mild impaired renal function: ≥90mL/min/1.73 m2
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG;
* Agree to take approved method of contraception during the clinical trail and 8 weeks after the last dose of apatinib. Female subject should be negative in the pregnancy test;

Exclusion Criteria:

for subjects with renal impairment

* Renal allograft recipients;
* Need hemodialysis during study;
* Uroclepsia or anuria;
* Allergic to apatinib or ingredients;
* History of heart disease in 12 months before study;
* Coagulation disorders;
* Hypertension and could not be controlled with hypotensor;
* With hepatic or archenteric disease;
* Participate in blood donation within 3 months before screening and donate blood volume ≥400mL, or receive blood transfusion, or donate blood volume≥200mL within 1 month prior dosing.
* Take any clinical trial drugs within 3 months prior dosing;
* Take any drugs that have effect on gastric acid and metabolic enzyme CYP 3A in 14 days before dosing;
* Addicted to alcohol and tobacco, drinking 14 units of alcohol per week (1 unit = 285 mL of beer, or 100mL of wine), or take ≥5 cigarettes;
* Positive in urine drug test;
* Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection;
* Anyone who refuse to stop ingesting drinks containing methylxanthine, or grapefruit or grapefruit-containing products from 48 hours before dosing to the end of the study;
* The investigator believes that the subjects are not eligible to participate in this trial.

for healthy subjects:

* Renal allograft recipients;
* Allergic to apatinib or ingredients;
* History of heart disease in 12 months before study;
* Coagulation disorders;
* Hypertension and could not be controlled with hypotensor;
* With hepatic or archenteric disease;
* Participate in blood donation within 3 months before screening and donate blood volume ≥400mL, or receive blood transfusion, or donate blood volume≥200mL within 1 month prior dosing.
* Take any clinical trial drugs within 3 months prior dosing;
* Take any drugs that have effect on gastric acid and metabolic enzyme CYP 3A in 14 days before dosing;
* Addicted to alcohol and tobacco, drinking 14 units of alcohol per week (1 unit =285 mL of beer, or 100mL of wine), or take ≥5 cigarettes;
* Positive in urine drug test;
* Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection;
* Anyone who refuse to stop ingesting drinks containing methylxanthine, or grapefruit or grapefruit-containing products from 48 hours before dosing to the end of the study;
* The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0-96 hours
  Maximum plasma concentration
AUC0-t | 0-96 hours
  Area under the plasma concentration versus time curve from zero to 96h
AUC0-∞ | 0-96 hours
  Area under the plasma concentration versus time curve from zero to infinity